CLINICAL TRIAL: NCT07314827
Title: A Feasibility Study Examining the Comparison of Transcendental Meditation Versus Health Education on Psychological and Hemodynamic Function in Post-menopausal Women
Brief Title: Women's Healthy Aging and Menopause; (WHAM)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, E. Robert Schwartz, Professor and Chair Emeritus, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20250622
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Meditation; Health Education
MeSH Terms: conditions — Health Education | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcendental Meditation (TM) (Experimental): Participants receive a standardized Transcendental Meditation (TM) program delivered over 12 weeks by a certified instructor, including orientation, structured instruction, follow-up seminars, and daily home practice.
  Interventions: Behavioral: Transcendental Meditation (TM)
- Women's Health Education (WHE) (Active Comparator): Participants receive a structured health education program over 12 weeks focused on menopause and cardiovascular health, delivered via Zoom and WhatsApp using evidence-based materials.
  Interventions: Behavioral: Women's Health Education (WHE)

INTERVENTIONS:
Behavioral: Transcendental Meditation (TM) — Orientation: 18-minute self-guided video; 30-45 minute remote group introductory talk.
  Instructional phase: 10-minute individual interview (phone/Zoom); one 60-75 minute in-person 1:1 TM instruction session at Miami TM Center, Lennar Center, or University of Miami (UM) Osher Center; three consecutive in-person group sessions (60-75 minutes each).
  Follow-up seminars: Six sessions over nine weeks (in person or Zoom), including a "10th Day Check" and additional ~30-minute seminars at 1, 2, and 3 months.
  Home practice: Two daily TM sessions (20 minutes each, morning and evening).
  Arms: Transcendental Meditation (TM)
Behavioral: Women's Health Education (WHE) — Stage 1: 30-minute video and introductory lecture on menopause and cardiovascular health.
  Stage 2: 60-minute one-on-one health coach meeting plus nutrition video. Stage 3: Eight sessions (~30 minutes each) with health check-ins, materials, and videos covering physical activity for heart and bone health, sleep and stress management during menopause, and lifestyle goal review and planning.
  Arms: Women's Health Education (WHE)

SUMMARY:
The present study will examine whether women at high risk for developing hypertension, i.e., post-menopausal status, at least mild psychological distress, and mildly elevated blood pressure, show improvements in these risk factors after a 12-week Transcendental Meditation (TM) intervention compared to Women's Health Education (WHE). Positive findings will provide initial evidence of using nonpharmacological methods, such as TM, to prevent hypertension in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. ≥130 systolic blood pressure (SBP) ≤160 and/or 84 ≥ diastolic blood pressure (DBP) ≤100.
2. Perceived stress scale (PSS-4) > 5
3. Able to give informed consent.
4. Understand study procedures and comply with them for the length of the study.
5. Ages between 50 and 80 years.
6. Post-menopausal ≥ 1 year since last menstruation
7. Reads and speaks English
8. UHealth patients
9. Working at least part-time

Exclusion Criteria:

1. Currently in a meditation program.
2. Meditates more than once per week
3. Recent stroke or cerebral neurologic impairment.
4. Current uses of mood stabilizers or antipsychotics.
5. Has been diagnosed with bipolar disorder, schizophrenia, or substance use disorder.
6. Inability to give written informed consent in English.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will only enroll only female participants because we are looking at the relationship between menopause and blood pressure.
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility-The number of individuals approached vs participate. | up to 3 years
  Recruiters will record the numbers of individuals who agree to participate vs interested in hearing about the study.
Recruitment feasibility-Reasons for not participating | up to 3 years
  A checklist completed by recruiters (schedule, time commitment, topic, ineligible, other)
Attendance feasibility - Training sessions attended by TM and WHE group | 12 weeks
  Training sessions attended by the TM participants as well as the attendance and participation in videos watched for the WHE group will be recorded.
Compliance feasibility - The number of meditation sessions per week for the TM participants. | 12 and 24 weeks
  Participants in the TM group estimate in the last month how many days per week they meditated (0 = not at all, 1 = up to 3 days per week, 2 = nearly every day once per day, 3 = nearly every day twice per day)
Stress - Perceived Stress Scale-10 (PSS-10) | Baseline, 8, 12, and 24 weeks
  Validated self-reporting instrument with 10 questions on perceived stress. Each question is rated on a 5-point Likert scale ranging from 0 = never to 4 = Very Often, referring to experiences in the past month. Total scores range from 0 to 40, higher = more stress.
Depressed mood - Patient Health Questionnaire-9, (PHQ-9) | Baseline, 8, 12, and 24 weeks
  A 9-item self-report measure of depressive symptoms. Each question is rated on a scale of 0 to 3, based on how often the symptom has been experienced in the past two weeks (0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day). The total score ranges from 0 to 27, higher scores indicating more severe depression.
Anxiety - Generalized Anxiety Disorder-7, (GAD-7) | Baseline, 8, 12, and 24 weeks
  A 7-item self-report questionnaire assessing symptoms of generalized anxiety disorder. Items are rated on a scale of 0-3 based on frequency over the past two weeks (0 = Not at all, 1 = Several days, 2 = More than half the days, 3 = Nearly every day). The total score ranges from 0-21, with higher scores indicating more severe anxiety symptoms.
Pain - Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference and Pain Intensity | Baseline, 8, 12, and 24 weeks
  Patient-reported outcomes from the PROMIS system. Pain Interference items assess the extent to which pain hampers daily activities, social, and emotional functioning. Pain Intensity is assessed with a 0-10 numeric rating scale for worst, average, and current pain. Higher scores indicate greater pain burden.
Menopausal Symptoms - Greene Climacteric Scale (GCS) | Baseline, 8, 12, and 24 weeks
  A 21-item questionnaire assessing menopausal symptoms across four domains: psychological (anxiety/depression), somatic (aches, headaches), vasomotor (hot flashes, night sweats), and sexual function. Each item is scored 0-3 (0 = Not at all, 3 = Extremely). Total and subscale scores indicate severity of menopausal symptoms.
Fruits and Vegetables Intake | Baseline, 8, 12, and 24 weeks
  A brief dietary assessment asking participants to report the average number of daily servings of fruits and vegetables consumed. Responses are recorded as number of servings per day.
24-hour Hemodynamic Monitoring | Baseline and 12 weeks
  Continuous ambulatory monitoring using Bio-Beat patches and a Polar chest strap. Measures include systolic and diastolic blood pressure, and heart rate averaged over 24 hours. Provides objective cardiovascular data.

SECONDARY OUTCOMES:
Acceptability quantitative - Satisfaction with interventions | 12-weeks post interventions
  Satisfaction with interventions Likert Scale (0-4, with 0 as not at all satisfied and 4 as extremely satisfied).
Acceptability qualitative - Strengths and weaknesses of the interventions | 12-weeks post intervention
  Participants will be asked to write one to two sentences on the strengths and one to two sentences on the weaknesses of the intervention e.g., time commitment, travel to sites (TM group)
Mental Well-being - Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Baseline, 8, 12, and 24 weeks
  A 14-item self-report scale assessing positive mental health and well-being. Each item is rated on a 5-point Likert scale from 1 = None of the time to 5 = All of the time, based on experiences over the past two weeks. Total scores range from 14-70, with higher scores reflecting greater well-being.
Insomnia - Insomnia Severity Index (ISI) | Baseline, 8, 12, and 24 weeks
  A 7-item self-report measure assessing the nature, severity, and impact of insomnia. Each item is scored on a 0-4 scale (0 = No problem, 4 = Very severe problem) based on the previous two weeks. Total scores range from 0-28, with higher scores indicating more severe insomnia symptoms.
Primary Care Probable Post-Traumatic Stress Disorder (PTSD) Screen for Diagnostic and Statistical Manual for Mental Disorders (DSM-5) (PC-PTSD-5) | Baseline, 8, 12, and 24 weeks
  A 5-item self-report screening tool for post-traumatic stress disorder. Respondents indicate whether they have been bothered by PTSD symptoms in the past month with a yes/no format. A cutoff of 3 or more positive responses suggests probable PTSD.
Brief Resilience Scale (BRS) | Baseline, 8, 12, and 24 weeks
  A 6-item self-report questionnaire assessing the ability to bounce back or recover from stress. Each item is rated on a 5-point scale from 1 = Strongly disagree to 5 = Strongly agree. Scores are averaged, with higher scores reflecting greater resilience.
Leisure Time Exercise Questionnaire (LTEQ) | Baseline, 8, 12, and 24 weeks
  A self-report questionnaire measuring the frequency of mild, moderate, and strenuous exercise during free time in a typical week. Frequencies are weighted by estimated metabolic equivalents (METs) and summed to yield a total exercise score.
Health Status and Medications | Baseline, 8, 12, and 24 weeks
  Participants self-report current health status and provide details on prescribed medications, including type, dosage, and frequency. This measure tracks changes in medication use over time.

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Schwartz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No